CLINICAL TRIAL: NCT06623292
Title: The Effect of Motivational Interviewing-Based Breastfeeding Education Given to Mothers With Infants in the Neonatal Intensive Care Unit on Breastfeeding Motivation and Breastfeeding Self-Efficacy: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing-Based Breastfeeding Education on Breastfeeding Motivation and Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 26.04.2024-04/05
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Breastfeeding; Motivation; Self Efficacy
Keywords: Breastfeeding motivation; Breastfeeding self-efficacy; Motivational interview
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to experimental and control groups using block randomization method. Randomization of mothers will be done according to maternal age and number of births. Maternal age (19-25 years and 26 years and older) and number of births (primiparous and multiparous) variables will be used for block randomization. In order to reach the sample size calculated in the study, strata will be repeated six times (2X2X6) and 24 mothers will be included in each group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Mothers in this group will not receive any treatment in the study. Mothers will fill out the "Breastfeeding Self-Efficacy Scale" and "Breastfeeding Motivation Scale" four times: on the first day of the baby's NICU admission, when their baby is discharged, 15 days after discharge and one month later discharge. In addition, a follow-up form will be completed.
- Intervention group (Experimental): Mothers in this group will receive motivational interview-based breastfeeding education. Mothers will fill out the "Breastfeeding Self-Efficacy Scale" and the "Breastfeeding Motivation Scale" four times: on the first day of the baby's NICU admission, when their baby is discharged, 15 days after discharge and one month later discharge. In addition, a follow-up form will be completed.
  Interventions: Other: Motivational interviewing-based breastfeeding education

INTERVENTIONS:
Other: Motivational interviewing-based breastfeeding education — This program includes breastfeeding motivational interviewing consisting of a total of 4 sessions and breastfeeding education consisting of one session.
  Arms: Intervention group

SUMMARY:
This study is being conducted to examine the effect of a motivational interviewing-based breastfeeding education intervention provided to mothers whose infants are hospitalized in the neonatal intensive care unit on the mothers' breastfeeding motivation and breastfeeding self-efficacy.

DETAILED DESCRIPTION:
Midwives and nurses working in the Neonatal Intensive Care Unit (NICU) are in a unique position to support the breastfeeding process and breastfeeding self-efficacy of mothers whose babies are hospitalized in the NICU. Health care professionals can use a variety of methods to support mothers' breastfeeding self-efficacy and encourage breastfeeding. Individualized interventions, breastfeeding education, and motivational interviewing are some of them. Motivational interviewing is basically a client-centered psychosocial intervention that helps individuals discover and resolve ambivalent feelings about health behaviors, learn new skills, and improve existing skills. In the breastfeeding process, the mother's motivation and positive intention are shown to be important indicators of breastfeeding continuation.

Health education about breastfeeding provided by neonatal intensive care nurses to mothers whose babies are hospitalized in the NICU for various reasons is one of the important initiatives of nurses. The contribution of health education planned with effective educational techniques for both mother and baby is undoubtedly very valuable. However, one of the important variables that should not be forgotten in the success of this education provided by the nurse is motivation, which also affects the self-efficacy of mothers regarding breastfeeding. In order to ensure the readiness of mothers to be educated about the breastfeeding process and breastfeeding of the infant hospitalized in the NICU, it would be appropriate to support the health education planned for mothers whose infants are hospitalized in the NICU with a motivational interviewing intervention. Based on this information, the planned research will examine the effect of motivational interviewing-based breastfeeding education provided to mothers whose infants are hospitalized in the NICU on mothers' breastfeeding motivation and breastfeeding self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* A baby born at 38-42 weeks gestational week admitted to the NICU,
* Who started breastfeeding her baby in the NICU,
* Literate in Turkish,
* Open to communication and cooperation,
* Volunteered to participate in the study,
* Willing to breastfeed your baby,
* Have a smart phone and internet connection,
* Mothers who scored 60 or less on the Breastfeeding Self-Efficacy Scale in the pretest

Exclusion Criteria:

* Any chronic illness and pregnancy complications,
* A condition that prevents breastfeeding,
* The mother has a diagnosed psychiatric illness,
* Mothers with a history of substance abuse.
* The presence of an obstacle to oral feeding and sucking in the infant,
* The baby has genetic, congenital anomalies, neurological, cardiac and metabolic diseases,
* The baby has undergone surgery.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale-Short Form | On the first day of the baby's admission to the NICU (pretest), at discharge, 15 days after discharge, one month after discharge
  The scale is 5-point Likert type. The items of the scale are scored as 1= "I am never sure" and 5 = "I am always sure". All items of the scale are positive. The lowest score is 14 and the highest score is 70. An increase in scale scores indicates an increase in breastfeeding self-efficacy.
Breastfeeding Motivation Scale | On the first day of the baby's admission to the NICU (pretest), at discharge, 15 days after discharge, one month after discharge
  The scale has a 4-point Likert-type scale scoring system. Each item is scored between 1="Strongly Disagree" and 4="Strongly Agree". The score of the sub-dimensions is calculated by averaging the scale sub-dimension scores [136]. As the score obtained from the sub-dimension of the scale increases, the motivation representing the sub-dimension also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Study Chair — Istanbul Medeniyet University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University, Kadıköy, Istanbul
  - Istanbul Medeniyet University, Istanbul, Kadıköy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: July through December of 2025
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Addicks SH, McNeil DW. Randomized Controlled Trial of Motivational Interviewing to Support Breastfeeding Among Appalachian Women. J Obstet Gynecol Neonatal Nurs. 2019 Jul;48(4):418-432. doi: 10.1016/j.jogn.2019.05.003. Epub 2019 Jun 7. PMID 31181186
- [Background] Franco-Antonio C, Calderon-Garcia JF, Santano-Mogena E, Rico-Martin S, Cordovilla-Guardia S. Effectiveness of a brief motivational intervention to increase the breastfeeding duration in the first 6 months postpartum: Randomized controlled trial. J Adv Nurs. 2020 Mar;76(3):888-902. doi: 10.1111/jan.14274. Epub 2019 Dec 18. PMID 31782535